Phase II multicenter clinical trial to evaluate the efficacy and safety of ibrutinib in combination with rituximab, gemcitabine, oxaliplatin, and dexamethasone followed by ibrutinib as maintenance treatment in patients with diffuse large B-cell lymphoma refractory to the treatment or relapsing, non-candidates to receive a TACM.

### STATISTICAL ANALYSIS REPORT

26th of April 2021 (version 1.0)

### TITLE

Phase II multicenter clinical trial to evaluate the efficacy and safety of ibrutinib in combination with rituximab, gemcitabine, oxaliplatin, and dexamethasone followed by ibrutinib as maintenance treatment in patients with diffuse large B-cell lymphoma refractory to the treatment or relapsing, non-candidates to receive a TACM.

| SPONSOR | |
|------------------|---------|
| COORDINATORS | |
| MONITORING ORFAN | ISATION |

## INDEX

| LIST | OF ABBREVIATIONS 7 | |
|---|---|---|
| 1. D | EFINITIONS | 9 |
| 1.1 | POPULATIONS FOR ANALYSIS | 9 |
| 1.2 | EFFICACY ANALYSIS | 9 |
| 2. R | ESULTS 1 | 10 |
| 2.1 | POPULATIONS | 10 |
| | 2.1.1. Patients registered in the eCRF | 10 |
| | 2.1.2. Analyzable patients | 11 |
| | 2.1.3. Analysis populations | 12 |
| 2.2 | | 12 |
| | 2.2.1. Vital signs | 13 |
| 2.3 | | 15 |
| | 31 | 16 |
| | 2.3.2. Diagnosis: Other histological data | 17 |
| | 2.3.3. Current lymphoma exploration | 18 |
| | 2.3.4. Current stage: Rebiopsy and other current results | 20 |
| | 2.3.5. Current histology: diagnosis and agreement | 21 |
| | 2.3.6. Current Immunohistochemistry: diagnosis and agreement | 22 |
| | 2.3.7. Global diagnosis | 23 |
| 2.4 | PREVIOUS TREATMENTS LYMPHOMA | 25 |
| | | 28 |
| | | 28<br>22 |
| | | 29<br>32 |
| 2.0 | | <b>32</b><br>32 |
| | | 32 |
| | | 32 |
| | | 33 |
| | | 33 |
| | | 33 |
| 2.0 | | |
| 2.9 | | <b>35</b><br>35 |
| | | 35 |
| | | 36 |
| 2.1 | | 39 |
| 2.1 | | 33<br>41 |
| | | - |

| | 2.12. EF | FFICACY: RESPONSE | 42 |
|---|---|---|---|
| | 2.12.1.<br>TREATE | SUMMARY RESPONSE AT 4TH CYCLE AND AFTER INDUCTION IN PATIENTS | ۷<br>42 |
| | 2.12.2. | RESPONSE AT 4TH CYCLE IN TREATED PATIENTS | 43 |
| | 2.12.3.<br>RESPOI | RESPONSE AT 4TH CYCLE IN PATIENTS FROM AVAILABLE NSE POPULATION | 44 |
| | 2.12.4. | RESPONSE AT 6-8TH CYCLE IN TREATED PATIENTS | 45 |
| | 2.12.5.<br>RESPO | RESPONSE AT 6-8TH CYCLE IN PATIENTS FROM AVAILABLE NSE POPULATION | 46 |
| | 2.12.1. | ORR IN TREATED PATIENTS | 47 |
| | 2.12.2. | ORR IN PATIENTS FROM AVAILABLE RESPONSE POPULATION | 48 |
| | 2.13. EF | FICACY: SURVIVAL | 49 |
| | 2.13.1. | OVERALL SUVIVAL IN TREATED PATIENTS | 49 |
| | 2.13.1. | OVERALL SUVIVAL IN AVAILABLE RESPONSE POPULATION | 52 |
| | 2.13.2. | PROGRESSION FREE SURVIVAL IN TREATED PATIENTS | 55 |
| | 2.13.3.<br>POPULA | PROGRESSION FREE SURVIVAL IN AVAILABLE RESPONSE<br>ATION | 58 |
| | 2.13.4. | EVENT FREE SURVIVAL IN TREATED PATIENTS | 61 |
| | 2.13.5. | RESPONSE DURATION IN TREATED PATIENTS | 64 |
| | 2.13.1. | COMPLETE RESPONSE DURATION IN TREATED PATIENTS | 66 |
| | 2.13.2. | PARTIAL RESPONSE DURATION IN TREATED PATIENTS | 68 |
| | 2.13.3. | RESPONSE DURATION IN AVAILABLE RESPONSE POPULATION | 70 |
| | 2.14. SA | AFETY: TOXICITY | 71 |
| | 2.14.1. | MOST FREQUENT ADVERSE EVENTS AND TOXICITIES | 72 |
| | 2.14.1. | HEMATOLOGICAL AND NON-HEMTOLOGICAL TOXICITIES | 74 |
| | 2.14.1. | SAES | 78 |
| 3. | ANNEXES | | 81 |
| | 3.1. ANNEX | 1: RELEVANT PREVIOUS EVENTS | 81 |
| | | 2: PREVIOUS MEDICATION | 85 |
| | 33 VNNEA | 3: ALL TOYICITIES | 22 |

### LIST OF ABBREVIATIONS

AbbreviationsTerm explanationAEAdverse EventCRComplete responseeCRFCase Report Form

ECOG Eastern Cooperative Oncology Group

EFS Event Free Survival

GEL/TAMO Grupo Español de Linfoma/Trasplante Autólogo de Médula Ósea

HLA Human Leukocyte Antigen

LDCBG Linfoma difuso de células B grandes

LNH Linfoma no Hodgkin

NA Not aplicable ND Not Done

OR Overall Response
OS Overall survival

PET Positron Emission Tomography

PR Partial Response
PD Progression disease
PFS Progression Free Survival

R-GEMOX Rituximab-GEMOX SAE Serious Adverse Event

SD Stable Disease UK Unknown

### 1. DEFINITIONS

#### 1.1. POPULATIONS FOR ANALYSIS

The analysis populations are defined as:

- **Population of all treated patients**: defined as all patients receiving at least 1 dose of study drug.
- **Population with evaluable response**: defined as all patients with measurable disease at baseline, receiving at least 1 dose of study drug, and having at least 1 adequate post-baseline disease evaluation. An adequate disease assessment is defined as having sufficient evidence to correctly indicate whether or not disease progression has occurred. Patients who have died from progression are also considered to have had an adequate evaluation.
- **Safety population:** defined as all patients receiving at least 1 dose of study drug, which is the same definition as for the population of all treated patients.

#### 1.2. EFFICACY ANALYSIS

**Efficacy analysis:** final analysis of the primary endpoint, ORR (CR + PR) after 4 cycles, can be carried out 4 months after the last patient was enrolled, and will be based on the population of all treated patients. Response rates with confidence intervals (95% interval) will be presented. The TRG will be evaluated in accordance with local and centralized PET / CT evaluations.

Overall survival, PFS, event-free survival, and duration of response are defined as follows (Cheson et al., 2007):

**Overall survival (OS):** defined as the time between entry into the trial and death from any cause. It will be analyzed using the Kaplan-Meier method. Data on patients withdrawn from the study or unavailable for follow-up will be censored on the date of the last contact.

**Progression-free survival (PFS).** It is defined as the time elapsed from the inclusion of the first patient in the study until the progression of the disease or death from any cause

**Event-free survival (EFS).** It is defined as the time elapsed from inclusion in the trial to lymphoma progression, treatment failure, or death from any cause. It will be analyzed using the Kaplan-Meier method.

**Duration of response.** It will be calculated from the date there is an indication of CR or PR to the date of disease recurrence or progression. It will be analyzed using the Kaplan-Meier method.

## 2. RESULTS

## 2.1. POPULATIONS

### 2.1.1. Patients registered in the eCRF

Table 1. Patients registered by hospital

| | able 1. Patients registered by | | 0/ |
|-------------------------|--------------------------------|---|----|
| | | N | % |
| Hospital<br><br> | | | |
| | Total | | |
| | Yes | | |
| Analyzable <sub>-</sub> | No | | |
| | Total | | |

### 2.1.2. Analyzable patients

Table 2. Not analyzable patients

| No. | Study Subject ID | Hospital | Reason |
|-----|------------------|----------|--------|

Table 3. Analyzable patient by hospital

| | | Analyzable | | | | | |
|----------|-------|------------|----|-----|---|----|------|
| | | | No | Yes | | To | otal |
| | | N | % | N | % | N | % |
| | | | | | · | | |
| | | _ | | | | | |
| Hospital | | _ | | | | | |
| | Total | | | | | | |

### 2.1.3. Analysis populations

**Table 4. Analysis population** 

| | - постольный разрами. | N | % |
|----------------------|---------------------------------------|---|---|
| Treated patient | Yes | | |
| population | Total | | |
| Available seemens | Yes | | |
| Available response | No | | |
| patient population - | Total | | |
| Reason considered | At least one post-baseline evaluation | | |
| response not | Death due to progression | | |
| available | Total | | |

Table 5. List of patients excluded from Available response patient population

| | Study<br>Subject ID | Hospital | Available response | Reason considered response available (or not) | Overall<br>survival | Reason of<br>Death | Specify reason of Death |
|---|---|---|---|---|---|---|---|
| 1 | | | | | | | |
| 2 | | | | | | | |
| 3 | | | | | | | |
| 4 | | • | | | | | |

### 2.2. BASELINE CHARACTERISTICS

Table 6. Gender

| | | N | % |
|-------------------|--------|---|---|
| | Male | | |
| Gender (Baseline) | Female | | |
| | Total | | |

Table 7. Age

| | N | Mean | SD | Median | Min | Max |
|-------------|---|------|----|--------|-----|-----|
| Age (years) | | | | | | |

### Vital signs

Table 8. Vital signs 1

| | N | Mean | SD | Median | Min | Max |
|---------------------------------|---|------|----|--------|-----|-----|
| Systolic blood pressure | | | | | | |
| (Baseline) | | | | | | |
| <b>Diastolic blood pressure</b> | | | | | | |
| (Baseline) | | | | | | |
| Temperature (Baseline) | | | | | | |
| Weight (Baseline) | | | | | | |
| Height (Baseline) | | | | | | |

Table 9. Vital signs 2

| | | N | % |
|-------------------------|-------|---|---|
| | 0 | | |
| ECOG (Baseline) | 1 | | |
| | 2 | | |
| | Total | | |
| | Yes | | |
| B symptoms (Baseline) | No | | |
| | Total | | |
| Pre-existing condition, | Yes | | |
| relevant signs or | No | | |
| symptoms (Baseline) | Total | | |

All relevant previous events are listed in ANNEX 1: RELEVANT PREVIOUS EVENTS (page 40), and the following table contains those events present in at least 5% of the patients.

Table 10. Most frequent relevant previous events (present in at least 5% of patients)

| | pationts) | |
|-----------------|-----------|---|
| | | N |
| Relevant | | |
| previous events | | |

**Table 11. Previous medication** 

| | | N | % |
|---------------------|-------|---|---|
| Drovious | Yes | | |
| Previous medication | No | | |
| medication | Total | | |

All previous medications are listed in ANNEX 2: PREVIOUS MEDICATION (page 40), and the following table contains those medications present in at least 5% of the patients.

Table 12. Most frequent previous medication (present in at least 5% of patients)

| Tubic IZ. I | most request provides incursation (prosent in at least 678 or patier | 110/ |
|---|---|---|
| | | N |
| Previous | | |
| medication | | |

## 2.3. DIAGNOSIS

Table 13. Time from diagnosis and age at diagnosis

| | N | Mean | SD | Median | Min | Max |
|------------------------------|---|------|----|--------|-----|-----|
| Time from diagnosis to study | | | | | | |
| inclusion (months) | | | | | | |
| Age at diagnosis | | · | • | | | |

Table 14. Local histological diagnosis, centralized and agreement

| lable 14. Local histological diagnosis, centralized and agreement | | | | |
|---|---|---|---|---|
| | | | N | % |
| Uistalagies subtype at | LDCBG w | ithout specification | | |
| Histological subtype at diagnosis, local | | Others <sup>1</sup> | | |
| (Baseline) | LDC | BG specified <sup>2</sup> | | |
| | | Total | | |
| 2: LDC | BG specified | LDCGB rich in T | | |
| | 1: Others | Follicular lymphoma | | |
| | | | N | % |
| | LDCBG w | ithout specification | | |
| Histological subtype at | | Others <sup>3</sup> | | |
| diagnosis, <u>centralized</u> | | NA | | |
| review (Baseline) | | ND | | |
| | | Total | | |
| | | CD5+ B lymphoma | | |
| | | Could not be | | |
| | | determined with | | |
| | 3: Others | submitted sample | | |
| | | MO cylinder biopsy | | |
| | | without evidence of | | |
| | | neoplastic infiltration | | |
| | | | N | % |
| | | No | | |
| Agreement in histology a | at diagnosis | Yes | | |
| | | Total | | |

Table 15. Patients without agreement in Histological type at diagnosis

| | Study<br>Subject<br>ID | Hospital | Diagnosis date<br>(Baseline) | Histological subtype at diagnosis, local (Baseline) | Histological subtype at diagnosis, centralized review (Baseline) | Agreement in histology at diagnosis |
|---|---|---|---|---|---|---|
| 1 | | | | | | |
| 2 | | | | | | |
| 3 | | | | | | |
| 4 | | | | | | |

## 1.1.1.Diagnosis: Immunohistochemical type of LDCBG

Table 16. Immunohistochemical type of LDCBG at diagnosis

| | | N | % |
|---|---|---|---|
| Income a blade about a d | no-CGB | | |
| Immunohistochemical - | Others | | |
| type at diagnosis,<br>local (Baseline) | UK | | |
| local (Basellile) | Total | | |
| _ | CGB | | |
| Immunohistochemical _ | no-CGB | | |
| type of LDCBG at | NA | | |
| diagnosis, centralized _ | ND | | |
| review (Baseline) | UK | | |
| | Total | | |
| _ | Non-CGB local and centralized | | |
| A | Non-CGB local and CGB centralized | | |
| Agreement in — immunohistochemical — | Non-CGB local and missing centralized | | |
| at diagnosis – | Missing local and centralized | | |
| at diagnosis – | Other local and missing centralized | | |
| | Total | | |
| Agreement in _ | Yes | | |
| immunohistochemical _ | No | | |
| at diagnosis | Total | | |

Table 17. Patients without agreement in Immunohistochemical type of LDCBG at diagnosis

| | Study<br>Subject<br>ID | Hospital | Diagnosis date<br>(Baseline) | Immunohistochemical agreement at diagnosis (Yes/No) | Immunohistochemical agreement at diagnosis |
|---|---|---|---|---|---|
| 1 | | | | | |
| 2 | | | | | |
| 3 | | | | | |
| 4 | | | | | |
| 5 | | | | | |

## 1.1.2. Diagnosis: Other histological data

Other histological data at diagnosis.

Table 18. Other histological data

| | | N | % |
|----------------------------------------|----------|---|---|
| | ABC | | |
| | Not done | | |
| Nanostring result at | NA | | |
| diagnosis (Baseline) | ND | | |
| | UK | | |
| | Total | | |
| | 1 | | |
| | II | | |
| Lymphoma stage at diagnosis (Baseline) | III | | |
| diagnosis (Baseline) | IV | | |
| | ND | | |

| | UK |
|---------------------|-----------|
| | Total |
| | 0 |
| | 1 |
| | 2 |
| ECOG diagnosis —— | 3 |
| (Baseline) —— | ND |
| | UK |
| | Total |
| | Normal |
| LDU et die enserie | Increased |
| LDH at diagnosis —— | ND |
| (Baseline) | UK |
| | Total |
| | 0-1 |
| | 2 |
| _ | 3 |
| IPI diagnosis | 4 |
| (Baseline) | 5 |
| | ND |
| | UK |
| | Total |

## 1.1.3. Current lymphoma exploration

Table 19. Current lymphoma exploration

| | · | N | % |
|---|---|---|---|
| | Yes | | |
| Adenopathy (Baseline) | No | | |
| | Total | | |
| Specify adapapathy | Example: Bilateral supraclavicular, Axillary, mediastinal, | | |
| Specify adenopathy (Baseline) | hilar | | |
| (Baselille) | Total | | |
| Hepatomegaly<br>(Baseline) | Yes | | |
| | No | | |
| (Baseille) | Total | | |
| Splanamagaly | Yes | | |
| Splenomegaly (Baseline) | No | | |
| (Baselille) | Total | | |
| Lymphomotous | Yes | | |
| Lymphomatous involvement (Baseline) | No | | |
| involvement (Basenne) | Total | | • |
| Specify Lymphomatous Example: Bone, liver and bone marrow | | | |
| involvement (Baseline) | Total | | |

### 1.1.4. Current stage: Rebiopsy and other current results

Table 20. Histological, molecular and current stage

| | groun, morocular una curront ctag | N | % |
|---|---|---|---|
| | Yes | | |
| Rebiopsy (Baseline) | No | | |
| | Total | | |
| | CGB | | |
| | ABC | | |
| Current nanostring recult | Not done | | |
| Current nanostring result (Baseline) | NA | | |
| (Daseille) | ND | | |
| | UK | | |
| | Total | | |
| | II | | |
| | III | | |
| Current lymphoma clinical | IV | | |
| stage (Baseline) | NA | | |
| | ND | | |
| | UK | | |
| | Total | | |
| | Yes | | |
| | No | | |
| Current Bone marrow biopsy - | NA | | - |
| histological affectation ———————————————————————————————————— | ND | | |
| (Daseille) | UK | | |
| | Total | | |
| | Yes | | |
| | No | | |
| Current cytometry involvement | NA | | |
| (Baseline) | ND | | |
| | UK | | |
| | Total | | |

### 1.1.5. Current histology: diagnosis and agreement

**Table 21. Current Histological subtype** 

| | | N | % |
|---|---|---|---|
| | LDCBG without specification | | |
| | LDCBG specified | | |
| Current, <u>local</u> histological subtype | NA | | |
| (Baseline) | ND | | |
| | UK | | |
| | Total | | |
| Specify other histological | Example: LDCBG gastric | | |
| subtypes current, local (Baseline) | Total | | |
| | LDCBG without specification | | |
| Current histological subtype, | Others | | · |
| <u>centralized review</u> (Baseline) | NA | | • |
| | ND | | |

| | UK |
|---|---|
| | Total |
| Specify <u>other</u> current histological subtypes, centralized review (Baseline) | Example: Lymphoma B of the marginal |
| | zone/Lymphoma B with plasmocellular |
| | differentiation |
| | Total |
| Current concordance in Histology | No |
| at diagnosis | Yes |
| | Total |

Table 22. Patients without agreement in current histology diagnosis

| Study<br>Subject<br>ID | Hospital | Current, local<br>histological subtype<br>(Baseline) | Specify other<br>histological<br>subtypes<br>current, local<br>(Baseline) | Current histological subtype, centralized review (Baseline) | Specify other current histological subtypes, centralized review (Baseline) |
|---|---|---|---|---|---|
| 1 | | | | | |
| 2 | | | | | |
| 3 | | | | | |

### 1.1.6. Current Immunohistochemistry: diagnosis and agreement

Table 23. Agreement current immunohistochemical diagnosis

| | | N | % |
|-------------------------------|--------|---|---|
| _ | no-CGB | | |
| Current | NA | | |
| immunohistochemical | ND | | |
| type, <u>local</u> (Baseline) | UK | | |
| | Total | | |
| _ | CGB | | |
| Immunohistochemical | no-CGB | | |
| type of current | NA | | |
| LDCBG, centralized | ND | | |
| review (Baseline) | UK | | |
| _ | Total | | |
| Current _ | No | | |
| immunohistochemical | Yes | | |
| agreement | Total | | |

Table 24. Patients without agreement in current immunohistochemical diagnosis

| | Study<br>Subject<br>ID | Hospital | Current<br>immunohistochemical<br>agreement | Current<br>immunohistochemical<br>type, local (Baseline) | Immunohistochemical<br>type of current<br>LDCBG, centralized<br>review (Baseline) |
|---|---|---|---|---|---|
| 1 | | | | | |
| 2 | | | | | |
| 3 | | | | | |
| 4 | | | | | |

### 1.1.7. Global diagnosis

Table 25. Agreement current immunohistochemical diagnosis

| | i da i e zer 7 kg. e e i i e i i e i i i i i i i i i i i | | |
|---|---|---|---|
| | | N | % |
| Global <u>local</u> | no-CGB | | |
| diagnosis | Total | | |
| | no-CGB | | |
| | CGB | | |
| Global | LDCBG without specification | | |
| centralized | Others: Follicular lymphoma, Lymphoma B with plasmocellular differentiation | | |
| diagnosis | ND | | |
| | UK | | |
| | Total | | |
| Global | No | | |
| | Yes | | |
| agreement | Total | | |

Table 26. Patients without agreement in current immunohistochemical diagnosis

| Study<br>Subject<br>ID | Hospital | Global local<br>diagnosis | Global centralized diagnosis |
|---|---|---|---|
| 1 | | | |
| 2 | | | |
| 3 | | | |

## 1.2. PREVIOUS TREATMENTS LYMPHOMA

Table 27. Number of previous treatment lines

| | | | | | | N | % |
|---|---|---|---|---|---|---|---|
| | | | 1 | | | | |
| Number of previous treatment lines | | | 2 | | | | |
| | | s | 3 | | | | |
| (Baseline) | | | 4 | | | | |
| | | | 5 | | | | |
| | | | Total | | | | |
| | N | Mean | SD | Media | an | Min | Max |
| Number of previous treatment lines (Baseline) | | | | | | | |

Table 28. Previous treatment: 1st line

| | | N | % |
|------------------------|------------------------------------------|---|---|
| _ | CR | | |
| | PR | | |
| Best response previous | SD | | |
| treatment line 1 | PD | | |
| (Baseline) | ND | | |
| | UK | | |
| | Total | | |
| | Yes | | |
| Relapse or previous | No | | |
| progression line 1 | NA | | |
| (Baseline) | ND | | |
| _ | Total | | |
| First line treatment _ | Example: R- CHOP, Rituximab, Splenectomy | | • |
| (Baseline) | Total | | |

Table 29. Previous treatment: 2<sup>nd</sup> line

| | | N | % |
|---------------------------|--------------------------|---|---|
| | CR | | |
| D | PR | | |
| Best response | SD | | |
| previous treatment line 2 | PD | | |
| (Baseline) | NA | | |
| | UK | | |
| | Total | | |
| Deleman | Yes | | |
| Relapse or previous | No | | |
| progression line | NA | | |
| 2 (Baseline) | UK | | |
| 2 (Dascille) | Total | | |
| Second line | NA | | |
| treatment | Example: R-ESHAP, R-DHAP | | |
| (Baseline) | Total | | |

Table 30. Previous treatment: 3<sup>rd</sup> line

| | | N | % |
|------------------|-----------------------------|---|---|
| | PR | | |
| Best response | SD | | |
| previous | PD | | |
| treatment line 3 | NA | | |
| (Baseline) | UK | | |
| | Total | | |
| Relapse or | Yes | | |
| previous | No | | |
| progression line | NA | | |
| 3 (Baseline) | Total | | |
| Third line | NA | | |
| treatment | Example: BeGEV + Transplant | | |
| (Baseline) | Total | | |

Table 31. Previous treatment: 4<sup>th</sup> line

| | | N | % |
|---|---|---|---|
| | PR | | |
| Post vosmonos provious | PD | | |
| Best response previous —— treatment line 4 (Baseline) —— | NA | | |
| treatment line 4 (Baseline) | UK | | |
| | Total | | |
| Relapse or previous | Yes | | |
| progression line 4 | NA | | |
| (Baseline) | Total | | |
| Founds line treatment | NA | | |
| Fourth line treatment —— | Example: Prednisone + Brentuximab | | |
| (Baseline) — | Total | | |

### 1.3. AUTOLOGOUS STEM CELL TRANSPLANT

Table 32. Autologous stem cell transplant

| | Table 32. Autologous Stelli Cell tralispiant | | |
|---|---|---|---|
| | | N | % |
| Atotwowowlowtotics | Yes | | |
| Autotransplantation (Receling) | No | | |
| (Baseline) —— | Total | | |
| | 1st CR | | |
| | 1st PR | | |
| Situation | 2nd CR | | |
| autotransplantation | 2nd PR | | |
| (Baseline) | Others | | |
| | NA | | |
| | Total | | |
| Specify other | Example: PD located in right axillar region | | |
| (Baseline) | Total | | |
| | CR | | |
| | PR | | |
| Best response —— | PD | | |
| autotransplantation —— (Baseline) —— | NA | | |
| (Daseille) | UK | | |
| | Total | | |

| | Example: 0, 3, 6, 9 |
|-----------------------------------|---------------------|
| Response duration(Baseline) | NA NA |
| | UK |
| | Total |
| Relapse or progression (Baseline) | Yes |
| | NA |
| | Total |

Table 33. Response duration (autologous stem cell transplant)

| | N | Mean | SD | Median | Min | Max |
|------------------------------|---|------|----|--------|-----|-----|
| Response duration (Baseline) | | | | | | |

## 1.4. ALEOGENIC TRANSPLANT HEMATOPOIETIC PROGENITORS

Table 34. Allogenic transplant hematopoietic progenitors

| | | <u> </u> | |
|---------------------------|-------|----------|---|
| | | N | % |
| Alletropoplent (Pacalina) | No | | |
| Allotransplant (Baseline) | Total | | |

### 1.5. EXTRANODAL AND NODAL AFFECTATION

#### **Table 35. Extranodal Affectation**

| | | N | % |
|---|---|---|---|
| Fortune and all offers to the second | Yes | | |
| Extranodal affectation | No | | |
| at diagnosis<br>(Baseline) | ND | | |
| (Basellile) - | Total | | |
| Locations sytropodolo | ND | | |
| Locations extranodals (Baseline) | Example: 0, 1, 2, 3 | | |
| (Daseille) | Total | | |
| Specify extranodal | Example: Bone, Lung, Bone marrow | | • |
| affectation (Baseline) | Total | | |

#### **Table 36. Nodal Affectation**

| | | N | % |
|---|---|---|---|
| Nodal | Yes | | |
| affectation at | No | | |
| diagnosis | ND | | |
| (Baseline) | Total | | |
| Nodal | ND | | |
| locations | Example: 0, 1, 2, 3 | | |
| (Baseline) | Total | | |
| Specify nodal | Example: Bilateral adrenal burky mass, Retroperitoneal | | |
| affectation<br>(Baseline) | Total | | |

### 1.6. BASELINE ANALYTICS

### 1.6.1. HEMOGRAM

Table 37. Baseline analytics: Hemogram

| | N | Mean | SD | Median | Min | Max |
|------------------------------|---|------|----|--------|-----|-----|
| Hemoglobin Value (Baseline) | | | | | | |
| Leukocytes Value (Baseline) | | | | | | |
| Lymphocytes Value (Baseline) | | | | | | |
| Monocytes Value (Baseline) | | | | | | |
| Eosinophils Value (Baseline) | | | | | | |
| Neutrophils Value (Baseline) | | | | | | |
| Platelets Value (Baseline) | · | | | | · | |

### 1.6.2. BIOCHEMISTRY

Table 38. Baseline analytics: Biochemistry

| | N | Mean | SD | Median | Min | Max |
|---|---|---|---|---|---|---|
| Creatinine Value (Baseline) | | | | | | |
| Urea Value (Baseline) | | | | | | |
| Urate Value (Baseline) | | | | | | |
| Sodium Value (Baseline) | | | | | | |
| Potassium Value (Baseline) | | | | | | |
| Calcium Value (Baseline) | | | | | | |
| Glucose Value (Baseline) | | | | | | |
| Protein Value (Baseline) | | | | | | |
| Albumin Value (Baseline) | | | | | | |
| LDH Value (Baseline) | | | | | | |
| Gamma globulin Value (Baseline) | | | | | | |
| Meta2-seric microglobulin Value (Baseline) | | | | | | |
| OSTP/ALT Value (Baseline) | | | | | | |
| OSOT/AST Value (Baseline) | | | | | | |
| FA Value (Baseline) | | | | | | |
| GGT Value (Baseline) | | | | | | |
| BIL Value (Baseline) | | | | | | |
| IgG Determination Value (Baseline) | | | | | · | |
| IgA Determination Value (Baseline) | | | | | | |
| IgM Determination Value (Baseline) | | | • | | | |

### 1.6.3. COAGULATION TEST

Table 39. Baseline analytics: Coagulation test

| | N | Mean | SD | Median | Min | Max |
|-----------------------------|---|------|----|--------|-----|-----|
| TTP Value (Baseline) | | | | | | |
| TP Value (Baseline) | | | | | | |
| Fibrinogen Value (Baseline) | | | | | | |

### 1.6.4. IPI

Table 40. Baseline analytics: IPI

| | U.D.10 101 Duo | | | | | |
|----------------|----------------|-------|----|--------|-----|-----|
| | | | | N | | % |
| | | 0 | | | | |
| | | 1 | | | | |
| | | 2 | | | | |
| IPI (Baseline) | | 3 | | | | |
| | | 4 | | | | |
| | | 5 | | | | |
| | | UK | | | | |
| | | Total | | | | |
| | N | Mean | SD | Median | Min | Max |
| IPI (Baseline) | | | | | | |

### 1.6.5. LYMPHOMA SITUATION

Table 41. Baseline analytics: Lymphoma situation

| | | N | % |
|---|---|---|---|
| | Partial Response | | |
| 0:44: | Refractory disease | | |
| Situation | Relapse early untreated (<1 year after diagnosis) | | |
| lymphoma<br>(Baseline) | Relapse late untreated | | |
| (Daseille) - | UK | | |
| | Total | | · |

### 1.6.6. SEROLOGY

Table 42. Baseline analytics: Serology

| | | N | % |
|-------------------|----------|---|---|
| HIV antibodies | Negative | | |
| (Baseline) | Total | | |
| | Positive | | |
| Hepatitis C | Negative | | |
| (Baseline) | UK | | |
| | Total | | |
| | Negative | | |
| RNA VHC | NA | | |
| (Baseline) | ND | | |
| (Daseille) | UK | | |
| | Total | | |
| | Positive | | |
| | Negative | | |
| HbsAg (Baseline) | NA | | |
| nusay (baselille) | ND | | |
| | UK | | |
| | Total | | |

| | Positive |
|------------------------|-------------------|
| Austi I IIaa | Negative |
| Anti Hbc<br>(Baseline) | ND |
| (Daseille) | UK |
| | Total |
| | Positive |
| Anti Uha | Negative |
| Anti Hbs<br>(Baseline) | ND ND |
| (Daseille) | UK |
| | Total |
| | Positive |
| | Negative Negative |
| DNA VHB | NA |
| (Baseline) | ND |
| | UK |
| | Total |

### 1.7. OTHER TESTS

### 1.7.1. OTHER TESTS: PREGNANCY

**Table 43. Other test: Pregnancy** 

| | | N | % |
|----------------------------------------|----------|---|---|
| | Negative | | |
| | NA | | |
| Pregnancy test at inclusion (Baseline) | ND | | |
| | UK | | |
| | Total | | _ |

### 1.7.2. OTHER TESTS: CARDIOLOGY TEST

Table 44. Other test: Cardiology test

| | Table 44. Other test. Caralology test | N | % |
|-------------------|---------------------------------------|---|----|
| | | N | 70 |
| | Without significative alterations | | |
| | Significative alterations | | |
| ECG at inclusion | NA | | |
| (Baseline) | ND | | |
| | UK | | |
| | Total | | |
| | Yes | | |
| Cardiac — | No | | |
| ventricular | NA | | |
| ejection fraction | ND | | |
| (Baseline) | UK | | |
| | Total | | |
| | Ecocardio | | |
| | MUGA | | |
| Technique FE — | NA | | |
| (Baseline) — | ND | | |
| | Total | | |
| Result FE | Normal | | |
| (Baseline) | Total | | |

### 1.7.3. OTHER TESTS: COMORBIDITIES QUESTIONNAIRE

Table 45. Comorbidities questionnaire: Item results

| | | N | % |
|---------------------------------------|---------------|---|---|
| | Yes | | |
| CRS-G comorbidity scale has been done | No | | |
| (Baseline) | Total | | |
| 11 41. (D 12 ) | Example: 0, 1 | | |
| Hearth (Baseline) | Total | | |
| Howards and the (Banadhas) | Example: 0, 1 | | |
| Hypertension (Baseline) | Total | | |
| Hamatan datia wa asalan (Basalina) | Example: 0, 1 | | |
| Hematopoietic vascular (Baseline) | Total | | |
| D 1 4 (D 11 ) | Example: 0, 1 | | |
| Respiratory (Baseline) | Total | | |
| <b>ADI</b> ( <b>D</b> ) | Example: 0, 1 | | |
| ORL (Baseline) | Total | | |
| | Example: 0, 1 | | |
| Upper GI apparatus (Baseline) | Total | | |
| | Example: 0, 1 | | |
| Lower GI apparatus (Baseline) | Total | | |
| | Example: 0, 1 | | |
| Liver (Baseline) | Total | | |
| D 1/D !! ) | Example: 0, 1 | | |
| Renal (Baseline) | Total | | |
| 0 '' ' 'D '' ' | Example: 0, 1 | | |
| Genitourinary (Baseline) | Total | | |
| 2 | Example: 0, 1 | | |
| Skeletal muscle (Baseline) | Total | | |
| | Example: 0, 1 | | |
| Nervous system (Baseline) | Total | | |
| Endocrine-metabolic system and breast | Example: 0, 1 | | |
| (Baseline) | Total | | |
| , , | Example: 0, 1 | | |
| Psychiatric problems (Baseline) | Total | | |
| | Yes | | |
| | No | | |
| GAH (Baseline) | NA NA | | |
| ( | ND | | |
| | Total | | |

Table 46. Comorbidities questionnaire: Scores

| | | N | % |
|---|---|---|---|
| Number of categories that have scored: of the total | Example: 0, 1 | | |
| of 14 categories, count those that have not received a score of 0 | Total | | |
| Total score (adding all the points) | ding all the points) Example: 0, 1 | | |
| Total score (adding all the points) | Total | | |
| Severity index (total score/number of categories | Example: 0, 1 | | |
| that have scored) | Total | | |

| Number of categories that have scored with a score>=3 | | Example: 0, 1 | | | | | |
|---|---|---|---|---|---|---|---|
| | | Total | | | | | |
| Number of categories that have scored with sco | | h score | Example: 0, 1 | | | | |
| 4 | 4 | | Total | | | | |
| | N | Mean | SD | Med | dian | Min | Max |
| Score > 0 (Baseline) | | | | | | | |
| Score (Baseline) | | | | | | | |
| Severity index (Baseline) | | | | | | | |

## 1.8. TREATMENT COMPLIANCE

| Table 47. Treatment compliance In | duction: Received | d cycles | com | plete | <u>d</u> |
|---|---|---|---|---|---|
| | | | N | | % |
| Number of induction cycles received - | Example: 1.00, 2 | .00 | | | |
| <u> </u> | Total | | | | |
| Number of induction cycles received _ | Example: 1.00, 2 | .00 | | | |
| complete (according to protocol) | Total | | | | |
| <u>_</u> | No | | | | |
| Patients with delayed induction cycles _ | Yes | | | | |
| | Total | | | | |
| % of induction cycles received complete | % of induction c | ycles | | | |
| (according to protocol) | received | | | | |
| , | Total | | | | |
| Number of induction cycles received | Example: 1.00, 2 | .00 | | | |
| with delay | Total | | | | |
| % of induction cycles received with | % of induction c | | | | |
| delay – | received with del | lay.00 | | | |
| • | Total | | | | |
| No official attended to the delication of the form | Not delayed cycle | | | | |
| No. of induction cycles delayed due to hematological toxicity | | | | | |
| hematological toxicity | Example: 1.00, 2<br>Total | .00 | | | |
| | N Mean SI | D Medi | an N | /lin | Max |
| Number of induction cycles received | | | - | | |
| Number of induction cycles received | | | | | |
| complete (according to protocol) | | | | | |
| % of induction cycles received complete | | | | | |
| (according to protocol) | | | | | |
| Number of induction cycles received with | | | | | |
| delay | | | | | |
| % of induction cycles received with delay | | | | | |
| No. of induction cycles delayed due to | | | | | |
| hematological toxicity | | | | | |
| Table 49 lbr | utinih dosago | | | | |
| Table 48. lbr | utinib dosage | NI NI | | | 0/_ |
| Table 48. lbr | | N | | | % |
| | 560mg/day | N | | | % |
| Minimum dose of ibrutinib received per | 560mg/day<br>420mg/day | N | | , | % |
| | 560mg/day<br>420mg/day<br>280mg/day | N | | | % |
| Minimum dose of ibrutinib received per | 560mg/day<br>420mg/day<br>280mg/day<br>Total | N | | , | % |
| Minimum dose of ibrutinib received per | 560mg/day<br>420mg/day<br>280mg/day | N | | | % |

### **Table 49. Treatment duration**

| | N | Mean | SD | Median | Min | Max |
|-----------------------------|---|------|----|--------|-----|-----|
| Treatment duration (months) | | | | | | |

### 1.9. END OF TREATMENT

Table 50. End of treatment

| | Table 50. Eliu of treatilient | | |
|---|---|---|---|
| | | N | % |
| Treatment ends Yes | | | |
| rreatment ends | Total | | |
| | Progression | | |
| | Unacceptable toxicity | | |
| Reason end of | End of maintenance | | |
| treatment (End of | Investigator criteria | | |
| treatment) | Patient withdrawal of continuing with treatment | | |
| | Others | | |
| | Total | | |
| Specify | Example: Allogeneic transplant, Cardiac | | |
| Other/Unacceptable | complications | | |
| toxicity or<br>Investigator criteria | Total | | |

### 1.10. EFFICACY: RESPONSE

1.10.1. SUMMARY RESPONSE AT 4TH CYCLE AND AFTER INDUCTION IN TREATED PATIENTS

Table 51. Summary of local response in the 4th cycle, 6-8th cycles in local evaluation (treated patients) and ORR

| | After 4th<br>cycle<br>N (%) | After induction N (%) | ORR (as<br>Best<br>Overall<br>Response) |
|---|---|---|---|
| Complete response (CR) | | | |
| Partial response (PR) | | | |
| Global response (GR=CR+PR) | | | |
| Stable disease (SD) | | | |
| Progression | | | |
| Not evaluated due to lack of follow-up at cycle 6-8 | | | |
| Not evaluated due to other reasons | | | |
| Total | | | |

### 1.10.2. RESPONSE AT 4TH CYCLE IN TREATED PATIENTS

Table 52. Response at 4th cycle in local evaluation (treated patients)

| | or our respective at this eyers in result or an author (in success p | utionito, |
|---|---|---|
| | | N (%, CI 95%) |
| | CR | |
| | PR | |
| Local | SD | |
| evaluation CT | Progression | |
| scan 4th cycle | Study ends due to Exitus without CT scan 4th cycle | |
| | Study ends due to IC withdrawal without CT scan 4th cycle | |
| | Total | |
| CR or PR at 4th | PR or CR | |
| cycle in local | No PR or CR | |
| evaluation | Total | |

Table 53. Response at 4th cycle in centralized evaluation (treated patients)

| iai | ne 33. Response at 4th cycle in centralized evaluation (treated | patients) |
|---|---|---|
| | | N (%, CI 95%) |
| | CR | |
| | PR | |
| Centralized | SD | |
| evaluation | Progression | |
| CT scan 4th | Study ends due to Exitus without CT scan 4th cycle | |
| cycle | Study ends due to IC withdrawal without CT scan 4th cycle | |
| | Without centralized response CT scan 4th cycle (local available) | |
| | Total | |
| CR or PR at | PR or CR | |
| 4th cycle in | No PR or CR | |
| centralized | Without centralized response CT scan 4th cycle (local available) | |
| evaluation | Total | |

## 1.10.3. RESPONSE AT 4TH CYCLE IN PATIENTS FROM AVAILABLE RESPONSE POPULATION

Table 54. Response at 4th cycle in local evaluation (evaluable assessment)

| Table 3 | i. Response at 4th cycle in local evaluation (evaluable assessment) |
|---|---|
| | N (%, CI 95%) |
| | CR |
| | PR |
| Local - | SD |
| evaluation CT —<br>scan 4th cycle —<br>— | Progression |
| | Study ends for Exitus without CT scan 4th cycle |
| | Total |
| CR or PR at 4th | PR or CR |
| cycle in local | No PR or CR |
| evaluation | Total |
| cycle in local | No PR or CR |

Table 55. Response at 4th cycle in centralized evaluation (evaluable assessment)

| | con response at him system continuing a system (system and system) | |
|---|---|---|
| | | N (%, CI 95%) |
| | CR | |
| | PR | |
| Centralized | SD | |
| evaluation | Progression | |
| CT scan 4th -<br>cycle - | Study ends for Exitus without CT scan 4th cycle | |
| | Without centralized response CT scan 4th cycle (local available) | |
| | Total | |
| CR or PR at | PR or CR | |
| th cycle in | No PR or CR | |
| centralized | Without centralized evaluation | |
| evaluation | Total | |

### 1.10.4. RESPONSE AT 6-8TH CYCLE IN TREATED PATIENTS

Table 56. Response at 6-8th cycle in local evaluation (treated patients)

| N (%, CI 95%) |
|---------------|

Table 57. Response at 6-8th cycle in centralized evaluation (treated patients)

| | | N (%, CI 95%) |
|---|---|---|
| | Positive* | |
| | Negative* | |
| | Progression in PET-TAC 4th cycle centralized (without evaluation | |
| Centralized | at 6-8th cycle) | |
| evaluation | Ends study due to Exitus without CT-scan 6-8th cycle | |
| CT scan | Ends study due to withdrawal of IC without CT-scan 6-8th cycle | |
| 6-8th cycle | Without CT-scan 6-8th cycle due to lack of follow-up | |
| | Without centralized evaluation 6-8th cycle (local available) | |
| | Without centralized evaluation 6-8th cycle | |
| | Total | |
| CR or PR at | Positive (Response)* | |
| 6-8th cycle in | Negative (No response)* | |
| centralized | Without CT scan at 6-8th | |
| evaluation | Total | 64 |

## 1.10.5. RESPONSE AT 6-8TH CYCLE IN PATIENTS FROM AVAILABLE RESPONSE POPULATION

Table 58. Response at 6-8th cycle in local evaluation (evaluable assessment)

| | | N (%, CI 95%) |
|---|---|---|
| | CR | |
| | PR | |
| Local — | SD | |
| evaluation — | Progression | |
| CT scan ——<br>6-8th cycle —— | Study ends for Exitus without CT scan 6-8th cycle | |
| | Without CT scan 6-8th cycle due to lack of follow-up | |
| | Total | |
| CR or PR at | PR or CR | |
| 6-8th cycle | No PR or CR | |
| in local | Without CT scan at 6-8th cycle due to lack of follow-up | |
| evaluation | Total | |

Table 59. Response at 6-8th cycle in centralized evaluation (evaluable assessment)

| assessment | |
|---|---|
| | N (%, CI 95%) |
| Positive* | |
| Negative* | |
| Progression in PET-TAC 4th cycle centralized (without evaluation | |
| at 6-8th cycle) | |
| Ends study due to Exitus without CT-scan 6-8th cycle | |
| Without CT-scan 6-8th cycle due to lack of follow-up | |
| Without centralized evaluation 6-8th cycle (local available) | |
| Without centralized evaluation 6-8th cycle | |
| Total | |
| Positive (Response)* | |
| Negative (No response)* | |
| Without CT scan at 6-8th | |
| Total | |
| | Positive* Negative* Progression in PET-TAC 4th cycle centralized (without evaluation at 6-8th cycle) Ends study due to Exitus without CT-scan 6-8th cycle Without CT-scan 6-8th cycle due to lack of follow-up Without centralized evaluation 6-8th cycle (local available) Without centralized evaluation 6-8th cycle Total Positive (Response)* Negative (No response)* |

### 1.1.1. ORR IN TREATED PATIENTS

Table 60. ORR in local evaluations (treated patients)

| | | N (%, CI 95%) |
|---|---|---|
| | CR | |
| | PR | |
| Daat Ownell | SD | |
| Best Overall | Relapse | |
| Response<br>(including<br>CT-scans after<br>EOT) | Progression | |
| | Study ends due to Exitus without CT scan 4th cycle and | |
| | after | |
| | Study ends due to IC withdrawal without CT scan 4th cycle | |
| | and after | |
| | Total | _ |

| BOR: CR or PR | No |
|---------------------|-------|
| (including | Yes |
| CT-scans after EOT) | Total |

### Table 61. ORR in centralized evaluations (treated patients)

| | | N (%, CI 95%) |
|---|---|---|
| BOR: CR or PR as | No | |
| Positive/Negative* (including CT-scans after EOT) centralized | Yes | |
| | Total | |

## 1.10.6. ORR IN PATIENTS FROM AVAILABLE RESPONSE POPULATION

### Table 62. ORR in local evaluations (evaluable assessment)

| | • | |
|---|---|---|
| | | N (%, CI 95%) |
| | CR | |
| D 1 O II | PR | |
| Best Overall | SD | |
| Response<br>(including | Relapse | |
| CT-scans after | Progression | |
| EOT) | Study ends due to Exitus without CT scan 4th cycle and | |
| LOT | after | |
| | Total | |
| BOR: CR or PR | No | |
| (including | Yes | |
| CT-scans after<br>EOT) | Total | |

### Table 63. ORR in centralized evaluations (evaluable assessment)

| | | N (%, CI 95%) |
|---------------------|-------|---------------|
| BOR: CR or PR as | No | |
| Positive/Negative* | V | |
| (including CT-scans | Yes | |
| after EOT) | Tatal | |
| centralized | Total | |

### 1.11. EFFICACY: SURVIVAL

### 1.11.1. OVERALL SUVIVAL IN TREATED PATIENTS

### Table 64. Overall survival in treated patients

| Estimated OS | N events | N at risk | % patients without exitus | CI 95% | % with exitu |
|---|---|---|---|---|---|
| at 6 months | | | | | |
| at 12 months | | | | | |
| at 24 months | | | | | |
| | N events (%) | Median | Min-Max | Standard error | CI 95% |
| Estimated OS | | | | | |

### Table 65. Overall survival in treated patients: Events and death reason

| | N (%; | CI 95%) |
|---|---|---|
| Overall | Alive | |
| Overall | Death | |
| survival | Total | |
| | Lymphoma/Progression | |
| D 41- | Toxicity | |
| Death | Others | |
| reason | Not specified | |
| | Total | |
| Specify de | leath | N (%) |
| reason | Example: CART-T therapy, Nosocomial respiratory infection | 1 |
| | Table 66. Follow-up time in treated patients | |

N Mea

N Mean (SE) Median (Min-Max)

Time until Death or last follow-up (from inclusion)

## 1.11.1.1 OVERALL SUVIVAL IN COMPLETE RESPONDERS (TREATED PATIENTS)

### Table 67. Overall survival in complete responders (treated patients)

| Estimated OS | N events | N at risk | % patients without<br>Death | CI 95% | % with Death |
|---|---|---|---|---|---|
| at 6 months | | | | | |
| at 12 months | | | | | |
| at 24 months | | | | | |
| | N events (%) | Median | Min-Max | Standard error | CI 95% |
| Estimated OS | | | | | |

Table 68. Overall survival in complete responders (treated patients): Events and death reason

| | | N (%; CI 95%) |
|---|---|---|
| Overell | Vivo | |
| Overall | Death | |
| survival | Total | |
| Danth | Lymphoma/Progression | |
| Death | Others | |
| reason | Total | |
| Specify de | eath | N (%) |
| reason | Example: Respiratory insufficiency due to p | progression |
| | Table 69. Follow-up time complete responders | (treated patients) |
| | N I | Mean (SE) Median (Min-Max) |
| Time unti | il exitus or last follow-up (from inclusion) | |

### 1.1.1. OVERALL SUVIVAL IN AVAILABLE RESPONSE POPULATION

| Tab | ole 70. Overall | survival ii | n available respo | nse populat | ion |
|---|---|---|---|---|---|
| Estimated OS | N events | N at risk | % patients without exitus | CI 95% | % with Death |
| at 6 months | | | | | |
| at 12 months | | | | | |
| at 24 months | | | | | |
| | N events (%) | Median | Min-Max | Standard<br>error | CI 95% |
| Estimated OS | | | | | |

Table 71. Overall survival in available response population: Events and death reason

| | | | N (%; CI 95%) |
|---|---|---|---|
| Occasil | Viv | 0 | |
| Overall survival | De | ath | |
| Survivai | To | al | |
| | Lyı | nphoma/Progression | |
| Death | Otl | ers | |
| reason | No | specified | |
| | Tot | al | |
| Specify do | ath | | N (%) |
| Specify de reason | auı | Example: CART-T therapy, Respiratory insufficiency progression | y due to |
| | | Table 72. Follow-up time in available response popu | lation |
| | | N Mean (S | E) Median (Min-Max) |
| Time unt | il exit | us or last follow-up (from inclusion) | _ |

# 1.1.1.1 OVERALL SUVIVAL IN COMPLETE RESPONDERS (AVAILABLE RESPONSE POPULATION)

Table 73. Overall survival in complete responders (available response population)

| | | PC | paiation | | |
|---|---|---|---|---|---|
| Estimated OS | N events | N at risk | % patients without exitus | CI 95% | % with exitus |
| at 6 months | | | | | |
| at 12 months | | | | | |
| at 24 months | | | | | |
| | N events (%) | Median | Min-Max | Standard error | CI 95% |
| Estimated OS | | | | | |

Table 74. Overall survival in complete responders (available response population): Events and death reason

| | | | N (%; CI 95%) |
|---|---|---|---|
| 0 | ۷i۱ | 70 | |
| Overall | De | ath | |
| survival | To | tal | |
| | Ly | mphoma/Progression | |
| Death | Ot | hers | |
| reason | To | tal | |
| | | | N (%) |
| Specify de reason | eath | Others: Probable septic shock with multi-organ failur (post-haploidentical transplantation) | e |
| | | Others: Respiratory insufficiency due to progression | |

Table 75. Follow-up time complete responders (available response population)

N Mean (SE) Median (Min-Max)

Time until exitus or last follow-up (from inclusion)

### 1.11.2. PROGRESSION FREE SURVIVAL IN TREATED PATIENTS

Table 76. Progression Free Survival in treated patients

| Estimated PFS | N events | N at risk | % of patients without PFS | CI 95% | % with PD |
|---|---|---|---|---|---|
| at 6 months | | | | | |
| at 12 months | | | | | |
| at 24 months | | | | | |
| | N (%) | Median | Min-Max | Standard<br>error | CI 95% |
| Estimated PFS | | | | | |

Table 77. PFS in treated patients: Events and PD assessment

| | | N (%; CI 95%) |
|-------------------------|---------------|---------------|
| | Vivo sin PD | |
| <b>Progression Free</b> | PD | |
| Survival | Death | |
| | Total | |
| DD accomment | | N (%) |
| PD assessment | PD assessment | |

## 1.11.2.1 PFS IN COMPLETE RESPONDERS (TREATED PATIENTS)

| Estimated PFS | N events | N at risk | % of patients without PFS | CI 95% | % with PD |
|---|---|---|---|---|---|
| at 6 months | | | | | |
| at 12 months | | | | | |
| at 24 months | | | | | |
| | N (%) | Median | Min-Max | Standard<br>error | CI 95% |
| Estimated PFS | | | | | |

| Table 79. PFS in | n complete responders (treated pat | ients): Events and PD assessment |
|---|---|---|
| | | N (%; CI 95%) |
| | Vivo sin PD | |
| <b>Progression Free</b> | PD | |
| Survival | Death | |
| | Total | |
| DD accomment | | N (%) |
| PD assessment | PD assessment | |
| | - | - |

## 1.11.3. PROGRESSION FREE SURVIVAL IN AVAILABLE RESPONSE POPULATION

Table 80. Progression Free Survival in available response population % of patients **Estimated PFS** N at risk CI 95% % with PD N events without PFS at 6 months at 12 months at 24 months Standard N (%) Median Min-Max CI 95% error **Estimated PFS** 

| Table 81. P | FS in available response population | n: Events and PD assessment |
|---|---|---|
| | | N (%; CI 95%) |
| | Vivo sin PD | |
| Progression Free<br>Survival | PD | |
| | Death | |
| | Total | |
| PD assessment | | N (%) |
| | PD assessment | |

## 1.11.3.1 PFS IN COMPLETE RESPONDERS (AVAILABLE RESPONSE POPULATION)

Table 82. Progression Free Survival in complete responders (available response population)

| Estimated PFS | N events | N at risk | % of patients without PFS | CI 95% | % with PD |
|---|---|---|---|---|---|
| at 6 months | | | | | |
| at 12 months | | | | | |
| at 24 months | | | | | |
| | N (%) | Median | Min-Max | Standard error | CI 95% |
| Estimated PFS | | | | | |

## Table 83. PFS in complete responders (available response population): Events and PD

| | assessillelli | |
|---------------------------|---------------|---------------|
| | | N (%; CI 95%) |
| | Vivo sin PD | |
| Progression Free Survival | PD | |
| | Death | |
| | Total | |
| DD accomment | | N (%) |
| PD assessment | PD assessment | |

### 1.11.4. EVENT FREE SURVIVAL IN TREATED PATIENTS

| Table | 84. | EFS | in | treated | l patients |
|-------|-----|-----|----|---------|------------|

| Estimated EFS | N events | N at risk | % patients without event | CI 95% | % patients with event |
|---|---|---|---|---|---|
| at 6 months | | | | | |
| at 12 months | | | | | |
| at 24months | | | | | |
| | N (%) | Median | Min-Max | Standard<br>error | CI 95% |
| Estimated EFS | | | | | |

### Table 85. EFS in treated patients: Events

| | | N (%; CI 95%) |
|----------------|--------------------------------|---------------|
| | Alive (without event) | |
| | PD | |
| Type of events | Death | |
| | Therapeutic failure (Toxicity) | |
| | Total | |

## 1.11.4.1 EFS IN COMPLETE RESPONDERS (AVAILABLE RESPONSE POPULATION)

Table 86. EFS in available response population

| Estimated EFS | N events | N at risk | % patients without event | CI 95% | % patients with event |
|---|---|---|---|---|---|
| at 6 months | | | | | |
| at 12 months | | | | | |
| at 24months | | | | | |
| | N (%) | Median | Min-Max | Standard<br>error | CI 95% |
| Estimated EFS | | | | | |

### Table 87. EFS in available response population: Events

| | | N (%; CI 95%) |
|----------------|--------------------------------|---------------|
| | Alive (without event) | |
| | PD | |
| Type of events | Death | |
| | Therapeutic failure (Toxicity) | |
| | Total | |

### 1.11.5. RESPONSE DURATION IN TREATED PATIENTS

### Table 88. TAC at which the CR or PR is reached (treated patients)

| | | N | % |
|---------------------|---------|---|---|
| TAC at which the CR | Cycle X | | |
| or PR is reached | Total | | |

### **Table 89. Response duration (treated patients)**

| • | N | Mean (SD) | Median (Min-Max) |
|-------------------------------------|---|-----------|------------------|
| Time since CR/PR until PD/exitus or | | | |
| censored | | | |

## 1.11.5.1 PFS FROM RESPONSE (CR or PR) IN TREATED PATIENTS

Table 90. PFS from response until PD/exitus (estimated by Kaplan-Meier) (in treated

| Estimated PFS from response | N events | N at risk | % of patients without event | CI 95% | % of patients with event |
|---|---|---|---|---|---|
| at 6 months | | | | | |
| at 12 months | | | | | |
| at 24 months | | | | | |
| | N (%) | Median | Min-Max | Standard error | CI 95% |
| Estimated PFS from response | | | | | |

#### Table 91. PFS from response (in treated patients): Events

| | • | 11 (0) 01 0 = 0 (1) |
|---------------------|----------------------------|---------------------|
| | | N (%; CI 95%) |
| | Alive without PD | |
| PFS from response | PD | |
| events | Exitus without previous PD | |
| | Total | |
| Dia with management | No | |
| Pts with response | Yes | |
| longer than 12m | Total | |

## 1.1.1.COMPLETE RESPONSE DURATION IN TREATED PATIENTS

#### Table 92. TAC at which the CR is reached (treated patients)

| | | N | % |
|---------------------|---------|---|---|
| TAC at which the CR | Cycle X | | |
| is reached | Total | | |

### Table 93. CR duration (treated patients)

| | | · / | |
|---|---|---|---|
| | N | Mean (SD) | Median (Min-Max) |
| Time since CR until PD/exitus or censored | | _ | |

## 1.1.1.1 PFS FROM <u>COMPLETE RESPONSE</u> IN TREATED PATIENTS

Table 94. PFS from CR until PD/exitus (estimated by Kaplan-Meier) (in treated patients)

| Estimated PFS from CR | N events | N at risk | % of patients without event | CI 95% | % of patients with<br>event |
|---|---|---|---|---|---|
| at 6 months | | | | | |
| at 12 months | | | | | |
| at 24 months | | | | | |
| | N (%) | Median | Min-Max | Standard<br>error | CI 95% |
| Estimated PFS from CR | | | | | |

Table 95. PFS from response (in treated patients): Events

| | | N (%; CI 95%) |
|--------------------|---------------------------|---------------|
| | Alive without PD | |
| PFS from CR | PD | |
| events | Death without previous PD | |
| | Total | |
| Dta with OD laws | No | |
| Pts with CR longer | Yes | |
| than 12m | Total | |

## PARTIAL RESPONSE DURATION IN TREATED PATIENTS

Table 96. TAC at which the PR is reached (treated patients)

| | | N | % |
|---------------------|---------|---|---|
| TAC at which the PR | Cycle X | | |
| is reached | Total | | |

Table 97. PR duration (treated patients)

| | 1 | | |
|-------------------------------------------|---|-----------|------------------|
| | N | Mean (SD) | Median (Min-Max) |
| Time since PR until PD/exitus or censored | | | |

## 1.1.1.2 PFS FROM <u>PARTIAL RESPONSE</u> IN TREATED PATIENTS

Table 98. PFS from PR until PD/exitus (estimated by Kaplan-Meier) (in treated patients)

| Estimated PFS from PR | N events | N at risk | % of patients without event | CI 95% | % of patients with event |
|---|---|---|---|---|---|
| at 6 months | | | | | |

| at 12 months | | | | | |
|---|---|---|---|---|---|
| at 24 months | | | | | |
| | N (%) | Median | Min-Max | Standard<br>error | CI 95% |
| Estimated PFS from PR | | | · | | |

| Table 99. PFS from response (in treated patients): Events | | |
|---|---|---|
| | | N (%; CI 95%) |
| DEC from DD | PD | |
| PFS from PR events | Death without previous PD | |
| events | Total | |
| Dto with DD longer | No | |
| Pts with PR longer than 12m | Yes | |
| ulali izili | Total | |

### 1.2. SAFETY: TOXICITY

As per protocol, the following definition is used to determine which adverse events are considered as toxicities:

### "Adverse event related to drug use

An adverse event is considered to be drug-related if the attribution is possible, probable, or very probable, based on the definitions provided below. (see page 54 of the protocol)".

| Table 10 | 0. Toxicities |
|----------------------------------|---------------|
| | N (%, IC 95%) |
| | No |
| AE | Yes |
| | Total |
| Toxicity: AE related to the | No |
| treatment (possible, probable or | Yes |
| definitively) | Total |
| | No |
| AE grade ≥3 | Yes |
| | Total |
| | No |
| Hematological Toxicity | Yes |
| | Total |
| | Yes |
| SAE | No |
| | Total |

#### 1.2.1. MOST FREQUENT ADVERSE EVENTS AND TOXICITIES

The following table shows the most frequent Adverse events taking a threshold of 5% and in overall and also taking into account the treatment phase at the date that the AEs first appeared.

Table 101. Most frequent AEs with 5% threshold

| • | Induction | Maintenance | Start day missing | Total |
|---|---|---|---|---|
| | N (%) | N (%) | N (%) | N (%) |
| Example: Platelet count decreased, Neutrophil count decreased | | | | |

The following table shows the most frequent <u>Toxicities</u> taking a threshold of 5% and in overall and also taking into account the treatment phase at the date that the AEs first appeared.

Table 102. Most frequent Toxicities with 5% threshold

| | Inductio | Maintenanc | Start day missing | Total |
|---|---|---|---|---|
| | n | е | Start day missing | Total |
| | N (%) | N (%) | N (%) | N (%) |
| Example: Diarrhea, Anemia | | | | |

The following table shows the most frequent <u>Toxicities</u> taking a threshold of 5%, according to their maximum grade in overall:

Table 103. Grades of most frequent Toxicities with 5% threshold. Overall

| | No | G-UK | G-1 | G-2 | G-3 | G-4 | Total |
|---|---|---|---|---|---|---|---|
| | N (%) | N (%) | N (%) | N (%) | N (%) | N (%) | N (%) |
| Example: Nausea, Anemia | | | | | | | |

Table 104. Grades of most frequent Toxicities (5% threshold), Induction phase.

| | No | G-UK | G-1 | G-2 | G-3 | G-4 | Total |
|---|---|---|---|---|---|---|---|
| | N (%) | N (%) | N (%) | N (%) | N (%) | N (%) | N (%) |
| Example: Nausea, Anemia | | | | | | | |

Table 105. Grades of most frequent Toxicities (5% threshold). Maintenance phase.

| | | No | G-UK | G-1 | G-2 | G-3 | G-4 | Total |
|----------|---------|-------|-------|-------|-------|-------|-------|-------|
| | | N (%) | N (%) | N (%) | N (%) | N (%) | N (%) | N (%) |
| Example: | Nausea, | | | | | | | |
| Anemia | | | | | | | | |

### 1.1.1. HEMATOLOGICAL AND NON-HEMTOLOGICAL TOXICITIES

The following table shows all the hematological toxicities (with maximum grade) taking into account the treatment phase at the date that the AEs first appeared.

Table 106. List of all hematological toxicities

| | Inductio<br>n | Maintenance | Total |
|---|---|---|---|
| | N (%) | N (%) | N (%) |
| Example: Anemia - Grade 1, Lymphocyte count decreased - Grade 2 | | | |

The following table shows all the non-haematological toxicities with maximum grade ≥3, taking into account the treatment phase at the date that the AEs first appeared.

**Table 107. List of non-hematological toxicities G≥3** 

| | Inductio | Maintenanc | Total |
|---|---|---|---|
| | n | е | IOtal |
| | N (%) | N (%) | N (%) |
| Example: Cefalea - Grade 3, Diarrhea - Grade 3 | | | |

The following table shows all the non-haematological toxicities with their maximum grades, taking into account the treatment phase at the date that the AE first appeared.

Table 108. List of non-hematological toxicities any grade

| | Induction | Maintenanc | AE<br>start<br>e day<br>missing | Total |
|---|---|---|---|---|
| | N (%) | N (%) | N (%) | N (%) |
| Example: Abdominal pain - Grade 2, Anorexia - Grade 2 | | | | |
| 1.1.1. SAES | | | | |
| Table 109. List of non-hematologic | al toxicities | G≥3 | | |
| | | Induction I | Maintenance | Total |
| | · | N (%) | N (%) | N (%) |
| Example: Abdominal pain - Grade 3, Anemia - Grade 3, Vomiting - Grade 3 | | | | |

| Study<br>Subject<br>ID | Hospital | AE with grade | Date AE start | Date AE end | Continuing at the end of study | AE related with<br>treatment (possible<br>/probable/<br>definitely) | Status | AEs according to treatment |
|---|---|---|---|---|---|---|---|---|

## 2. ANNEXES

### 2.1. ANNEX 1: RELEVANT PREVIOUS EVENTS

### Table 111. List of all relevant previous events

| | | N |
|---|---|---|
| Relevant previous events | Example: Arterial hypertension, Acute cholecystitis, Dyslipidemia | |

### 2.2. ANNEX 2: PREVIOUS MEDICATION

### Table 112. List of all previous medication

| | · | N |
|------------|--------------------------------------------|---|
| Previous | Example: Acetylsalicylic acid, Omeprazole, | |
| medication | Trimethoprim/sulfamethoxazole | |

## 2.3. ANNEX 3: ALL TOXICITIES

#### Table 113. List of all toxicities

| Study<br>Subjec<br>t ID | Hospital | AE with grade | Date AE start | Date AE<br>end | Continuing<br>at the end<br>of study | SAE | Status | Hematological<br>AE | AEs according to treatment |
|---|---|---|---|---|---|---|---|---|---|